CLINICAL TRIAL: NCT07064681
Title: The Real-World Study of Neoadjuvant Immune-Checkpoint Blockade Therapy Combining With TACE For Resectable Hepatocellular Carcinoma With High Recurrence Risk
Brief Title: The Real-world Study of AK104 Combining With TACE for Resectable Hepatocellular Carcinoma (MORNING)
Acronym: MORNING-RWS
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Professor, Sun Yat-sen University
Other Study IDs: RWS2024
Record Dates: First submitted 2025-07-05; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Resectable Hepatocellular Carcinoma With High Risk of Recurrence
Keywords: Resectable Hepatocellular Carcinoma with High Risk of Recurrence; Real-world study
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective group: retrospective group
  Interventions: Procedure: Surgery with and without the aid of Indocyanine Green (ICG)
- prospective group: prospective group
  Interventions: Procedure: Surgery with and without the aid of Indocyanine Green (ICG)

INTERVENTIONS:
Procedure: Surgery with and without the aid of Indocyanine Green (ICG) — Enrolled patients will receive surgery and be follow up for 2 years

SUMMARY:
This is an observational study. All patients who meet the inclusion criteria of our previous Phase 2, open-label, single-arm study of neoadjuvant immune-checkpoint blockade therapy (AK104) combining with TACE for resectable hepatocellular carcinoma, but refuse to receive neoadjuvant treatment will be asked again to participate this observational study retrospectively and prospectively. Participants will receive surgery and regular monitoring for 1 year. The purpose is to provide real-world cohort for comparison with the neoadjuvant cohort.

DETAILED DESCRIPTION:
This study will first retrospectively enroll the patients who meet the inclusion criteria of our previous neoadjuvant trial but refuse to receive neoadjuvant treatment. Then prospective enrollment will be taken following the same rules at the same of our neoadjuvant trial. Every enrolled patient will receive surgery without neoadjuvant therapy. Long-term survival follow-up will be conducted as well.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years but ≤75 years
2. Resectable HCC staged BCLC A/B
3. Treatment naïve for HCC
4. High risk for recurrence, meeting at least one of the following criteria:

   1. Multiple tumor lesions
   2. Individual tumor > 5cm
   3. AFP > 400 ug/L
   4. MVI positive based on preoperative MRI according to MVI predictive model of Radiomics
5. Measurable or evaluable lesions according to RECIST v1.1 criteria
6. ECOG performance status 0-1
7. Child-Pugh class A
8. Life expectancy ≥ 12 weeks
9. Adequate organ and marrow function as defined below:

   1. Hemoglobin ≥9.0 g/dL
   2. Absolute neutrophil count ≥ 1,500/μL
   3. Platelets count ≥ 75,000/μL
   4. Total serum bilirubin ≤ 1.5 ×upper limit of normal(ULN)
   5. AST and ALT ≤ 5 × ULN, ALP ≤ 4 ×ULN
   6. Serum creatinine ≤ 1.5 ×ULN
   7. INR ≤ 1.5 ×ULN, APTT ≤ 1.5 ×ULN
   8. Serum albumin ≥3.0 g/dL
10. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test.
11. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen as assessed by the treating investigator are eligible for this trial.
12. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Any prior treatment for HCC.
2. Tumor rupture or bleeding. Suspected abdominal metastasis.
3. A major surgical procedure, open biopsy, or significant traumatic injury with poorly healed wound within 6 weeks prior to enrollment.
4. History of allogenic organ transplantation.
5. Under other clinical trials.
6. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion: vitiligo or alopecia, hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement, any chronic skin condition that does not require systemic therapy or celiac disease controlled by diet alone.
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to AK104 or other immune checkpoint inhibitors.
8. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection (including tuberculosis), uncontrolled hypertension (defined as blood pressure of > 140/90 mmHg during the screening period despite medical management), interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs, or compromise the ability of the patient to give written informed consent.
9. History of hepatic encephalopathy, refractory ascites or esophagogastric varices with high risk of bleeding. Upper gastrointestinal hemorrhage within the year prior to the first dose of study drug.
10. Active hepatitis B infection without treatment (positive HBV surface antigen (HBsAg) and HBV DNA ≥ 1000 IU/ml). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Active hepatitis C infection (positive HCV antibody and HCV RNA above the lower limit of detection).
11. A primary brain tumor (excluding meningiomas and other benign lesions), any brain metastases, leptomeningeal disease, seizure disorders not controlled with standard medical therapy, or history of a stroke within the year prior to the first dose of study drug.
12. History of active primary immunodeficiency.
13. History of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
14. Current or prior use of immunosuppressive medication within 14 days prior to the first dose of study agent. The following are exceptions to this criterion: Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection). Systemic corticosteroids at physiologic doses that do not exceed 10 mg/day of prednisone or its equivalent. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
15. Receipt of live attenuated vaccine within 30 days prior to the first dose of study drug. Note: Patients, if enrolled, should not receive live vaccine whilst receiving study drug and for at least 30 days after the last dose of study agent.
16. Systemic immunostimulant therapy within 14 days prior to the first dose of study agent.
17. History of serious systemic disease, including myocardial infarction or unstable angina within the 12 months prior to the first dose of study drug, hypertensive crisis or hypertensive encephalopathy, New York Heart Association (NYHA) grade II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication, significant vascular disease or symptomatic peripheral vascular disease.
18. History of coagulopathy, bleeding diathesis, or thrombosis within the 12 months prior to the first dose of study drug.
19. A serious, non-healing wound, ulcer, or bone fracture.
20. Pregnancy or lactation.
21. Total parenteral nutrition.
22. Exclusion from the study by the judgement of investigators, due to some factors that may lead to the forced termination of the study, including other acute, chronic or psychological disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Resectable HCC patients with high risk of recurrence
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-05 (Estimated); Primary Completion 2025-12-17 (Estimated); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
1-year recurrence rate | 1-year recurrence rate
  1-year recurrence rate
1-year recurrence rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of SYSU, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided